CLINICAL TRIAL: NCT06675279
Title: The Headache Needs Assessment (HANA) Survey: Psychometric Properties of the Turkish Version in Migraine
Brief Title: Psychometric Properties of the Turkish Version of the HANA in Migraine
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Halime Arikan, Assistant Professor, Tokat Gaziosmanpasa University
Other Study IDs: 83116987-155
Record Dates: First submitted 2024-11-02; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-03

CONDITIONS: Migraine
Keywords: Headache Needs Assessment; Migraine; Turkish
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Individuals with migraine: The demographic information of individuals with migraines, along with data from the Visual Analog Scale, Migraine Disability Assessment Questionnaire, Headache Impact Test-6, Henry Ford Hospital Headache Disability Inventory, and Headache Needs Assessment, will be collected and analyzed.
  Interventions: Other: Survey-based study

INTERVENTIONS:
Other: Survey-based study — The demographic information of individuals with migraines, along with data from the Visual Analog Scale, Migraine Disability Assessment Questionnaire, Headache Impact Test, Henry Ford Hospital Headache Disability Inventory, and Headache Needs Assessment, will be collected and analyzed.

SUMMARY:
Migraine is one of the most common neurological disorders, affecting numerous adults. Headaches are often associated with significant disruptions that can interrupt the patient's usual activities for hours. Although headaches are typically episodic, many individuals with migraine experience life restrictions due to the anticipation of future attacks and the prevalent concern that headaches will compromise their functional capabilities. Several health-related quality of life scales have been developed to assess migraine and its associated conditions. Some examples include the Migraine-Specific Quality of Life Questionnaire, the Quality of Life and Migraine Scale, and the Migraine-Specific Quality of Life Measure. While some of these scales have Turkish versions, others do not. Many of these instruments are designed for clinical research, offering comprehensive assessment but are disadvantaged by lengthy completion and scoring times for patients. There is a need for brief health status measures with simple scoring systems that can evaluate the overall impact of migraines on daily activities. The Headache Needs Assessment (HANA) is a seven-item questionnaire developed to assess migraine-related quality of life issues.

This study aims to validate and establish the reliability of the Turkish version of the Headache Needs Assessment for evaluating individuals with migraines. If proven valid and reliable, the Headache Needs Assessment will be a practical tool for assessing the quality of life in individuals with migraines.

Null Hypothesis (H0): The Turkish version of the Headache Needs Assessment is not valid and reliable.

Alternative Hypothesis (H1): The Turkish version of the Headache Needs Assessment is valid and reliable.

DETAILED DESCRIPTION:
Migraine is a serious health problem that disrupts quality of life and ranks second among primary headaches, affecting over 10% of the general population. In Turkey, the lifetime prevalence of migraine is reported to be 16%, with rates of 10.9% in men and 21.8% in women. Migraine is characterized by episodic attacks that may include headaches accompanied by vomiting, nausea, phonophobia, or photophobia. Chronic migraine is defined as a headache occurring on 15 or more days per month for over three months, with migraine features present on at least 8 of those days. The International Classification of Headache Disorders criteria for migraine require only two of four commonly seen pain features; thus, a non-throbbing, bilateral headache can still meet migraine criteria if it is moderate to severe, worsens with physical activity, and is accompanied by migraine-specific symptoms. Neck pain related to stress, which is sometimes associated with tension-type headache, is also a common feature of migraine.

Measurements play a crucial role in scientific research across various fields, including natural sciences, social sciences, and health sciences. In the biomedical sciences, many clinical conditions, psychological behaviors, attitudes, and beliefs are challenging to measure accurately. These may include disease severity, disease-related quality of life, pain perception, anxiety, and more. To quantify and assess specific attributes, researchers develop tools known as "scales" that consist of various components. Clinical scales are tools used in medicine to evaluate different aspects of a patient's health, including physical and mental health symptoms, functional abilities, and overall quality of life.

The Headache Needs Assessment (HANA) is designed to assess two dimensions of the chronic impact of migraine-related quality of life issues: frequency and discomfort. It comprises seven items and serves as a useful screening tool for evaluating the impact of migraine on individuals. Its two-dimensional approach to patient-reported quality of life enables individuals to weigh the influence of both the frequency and discomfort of chronic migraines on various aspects of daily life. This scale will fill a gap in the Turkish literature regarding the parameters it evaluates and will serve as a valuable tool in the field.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of chronic migraine (headaches occurring on more than 15 days per month for over three months, with migraine headaches on at least eight days per month),
* Being between 18 and 65 years of age,
* Experiencing neck pain during migraine attacks.

Exclusion Criteria:

* Having a diagnosis of any headache disorder other than chronic migraine,
* Having a history of any systemic disease, such as malignancy, inflammatory conditions, acute fractures, surgical history, neurological, psychological, or rheumatological disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with migraine
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Headache Needs Assessment Survey | through study completion, an average of 6 months
  The Headache Needs Assessment consists of seven items that evaluate areas such as anxiety/worry, depression/discouragement, self-control, energy, functioning/work, family/social activities, and the overall impact of migraine. A distinctive feature of the questionnaire is that it separates responses into two categories: (1) How often did this issue occur? (1= Never, 2= Rarely, 3= Sometimes, 4= Often, 5= Always); and (2) How much did this issue bother you? (1= Not at all, 2= A little, 3= Somewhat, 4= Quite a bit, 5= Very much). The total score ranges from 14 to 70, with higher scores indicating a more negatively impacted quality of life.

SECONDARY OUTCOMES:
Visual Analog Scale | through study completion, an average of 6 months
  Headache severity was assessed using the Visual Analog Scale (VAS). A 10 cm horizontal line was drawn with a ruler for the VAS, where the beginning of the line (0 cm) was described to patients as "no pain," and the end of the line (10 cm) was described as "unbearable, severe pain." Patients were asked to mark a point on the line that best represented the intensity of their headache. The distance from the starting point to the marked point was then measured and recorded as the headache severity.
Migraine Disability Assessment Questionnaire | through study completion, an average of 6 months
  Disability related to migraines was assessed using the Migraine Disability Assessment Questionnaire (MIDAS). MIDAS evaluates disability over the past three months and consists of a five-item, self-administered test that addresses work/school-related disability, household chores, and family, social, or leisure activities. The total score is calculated based on the number of days missed in these activities, classifying disability as minimal (0-5 points), mild (6-10 points), moderate (11-20 points), or severe (≥21 points). The validity, reliability, and Turkish version of the questionnaire were established by Ertaş et al.
Headache Impact Test-6 | through study completion, an average of 6 months
  The Headache Impact Test-6 (HIT-6) is a quality of life questionnaire for headaches that evaluates vitality, pain, psychological distress, social functioning, role limitations, and cognitive functioning. Each item is scored on a 5-point Likert scale (6 = never, 8 = rarely, 10 = sometimes, 11 = very often, 13 = always). The total score is determined by summing the scores of all six items, ranging from 36 to 78. The scores are categorized as follows: ≤49 = little to no impact, 50-55 = some impact, 56-59 = substantial impact, and 60-78 = severe impact, with higher scores indicating greater impairment in quality of life. The validity, reliability, and Turkish version of the questionnaire have been established.
Henry Ford Hospital Headache Disability Inventory | through study completion, an average of 6 months
  The Henry Ford Hospital Headache Disability Inventory is a 25-item questionnaire that examines the impact of headaches on daily life. The inventory has a two-dimensional structure, comprising emotional and functional components. Each item is scored as No: 0, Sometimes: 2, and Yes: 4. The total score ranges from 0 to 100, with higher scores indicating greater headache-related disability. The validity, reliability, and Turkish version of the inventory were developed by Kılınç et al.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpaşa University, Tokat Province, Tokat Province, Turkey (Türkiye)